CLINICAL TRIAL: NCT00645138
Title: A Comparison of Ultrasound-assisted Paravertebral Block and General Anesthesia for Outpatient Breast Cancer Surgery, a Prospective Randomized Trial
Brief Title: Comparison of Paravertebral Block With General Anesthesia in Patients Undergoing Breast Cancer Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Tiffany Tedore MD, New York Presbyterian Hospital Weill Cornell Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0801009584
Record Dates: First submitted 2008-03-19; First posted 2008-03-27 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: breast carcinoma; breast cancer; paravertebral block; comparison of paravertebral block and general anesthesia; ultrasound
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paravertebral Block (Active Comparator): Patients receiving Paravertebral Block.
  Interventions: Procedure: Paravertebral Block
- General Anesthesia (Active Comparator): Patients receiving General Anesthesia.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Paravertebral Block — Sedation will be provided with midazolam and fentanyl. The transverse processes of T1-T6 will be located using ultrasound guidance. The area will be prepped with betadine. At each level, a 21 Gauge, 4-inch Stimuplex needle will be inserted in order to make contact with the transverse process. Once the transverse process has been located, the needle will be "walked off" the process and inserted 1 cm deep to its inferior border. After negative aspiration, 3 mL of 1.5% mepivacaine with epinephrine 1:200,000 and bicarbonate and 3 mL of 0.5% bupivacaine with epinephrine 1:200,000 will be injected. Sedation will be provided with 50-100 mcg/kg/min of propofol during the surgical procedure. Approximately 20 minutes before the end of the procedure, 4 mg of zofran will be administered.
  Arms: Paravertebral Block
Procedure: General Anesthesia — Patients in the general anesthesia group will receive midazolam preoperatively for anxiolysis. Anesthesia will be induced with propofol and fentanyl. An LMA will be inserted and anesthesia maintained with sevoflurane in air and oxygen. 4 mg of zofran will be administered approximately 20 minutes before the end of the surgical procedure. The LMA will be removed and the patient will be transported to the PACU at the conclusion of the surgery.
  Arms: General Anesthesia

SUMMARY:
The purpose of this project is to determine if there is a difference between paravertebral block and general anesthesia in terms of time to discharge from the Post-Anesthesia Care Unit and pain level in patients undergoing outpatient breast cancer surgery.

DETAILED DESCRIPTION:
The optimal anesthetic technique for breast cancer surgery allows for good postoperative pain relief and rapid discharge. Breast cancer surgery with potential axillary dissection is often performed under general anesthesia due to the potential for poor analgesia with local anesthetic infiltration at the surgical site alone. General anesthesia can be associated with increased post-operative pain, nausea, and delayed discharge when compared to regional anesthesia for breast and other types of procedures (1,2).

The paravertebral block is a technique that has been used perioperatively for breast (3,4), thoracic (5), abdominal (6), and hernia surgeries (7). It has also been used for pain control after rib fractures and penetrating trauma (8,9). The paravertebral block is performed by injecting local anesthetic above or below the transverse processes of the vertebral bodies where the spinal nerve roots emerge from the intervertebral foramina. The most common technique is to insert a needle 2.5 centimeters lateral to the spinous process at each level and "walk off" the transverse process. Injections at one or multiple levels block the somatic and sympathetic innervation to these dermatomes (10).

Rare complications of thoracic paravertebral blocks include epidural spread, intrathecal injection, and Horner's Syndrome (1,11,12). One of the most feared complications of the traditional technique is pleural puncture, which has an incidence of 0.64% to 6.7% in the published literature (3,11,13).

Ultrasound guidance in regional anesthesia is gaining widespread popularity. This technology provides visualization of key anatomic structures and has been shown to decrease block placement and onset times (14,15) and improve patient comfort (15). Ultrasound-guided blocks are associated with success rates of greater than 90% (15,16). In the thoracic region, ultrasound can be used to identify the vertebral transverse processes, as well as the ribs and the pleura of the lungs (17). In this way, pleural puncture can be avoided during paravertebral block placement.

To date there have been no published prospective, randomized trials comparing the multiple injection thoracic paravertebral technique using ultrasound guidance to general anesthesia in breast cancer surgery patients.

Our hypothesis is that paravertebral block anesthesia will result in shorter Post Anesthesia Care Unit (PACU) stays and decreased Visual Analog Scale (VAS) scores when compared to general anesthesia in patients undergoing breast cancer surgery. Secondary endpoints will include the need for postoperative opioids and the presence of nausea and/or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older with suspected breast carcinoma scheduled for unilateral lumpectomy or mass excision with sentinel node biopsy and possible axillary dissection.

Exclusion Criteria:

* A diagnosis of chronic pain, regular use of opioid medications, infection at the injection site, allergy to amide local anesthetics, bleeding disorder, contraindication to LMA, and patient refusal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Time in minutes until the patient is declared ready for discharge from the Post Anesthesia Care Unit (PACU) | Until PACU discharge
Visual Analog Scale (VAS) pain scores at 30, 60, 90, and 120 minutes after PACU admission. A VAS score will also be assessed on the first postoperative day. | Until PACU discharge and for 24 hours

SECONDARY OUTCOMES:
The need for postoperative opioids in the PACU and during the first postoperative day will be assessed. | 24 hours
Episodes of nausea or vomiting in the PACU and during the first postoperative day will be assessed. | 24 hours
Total time spent in the operating room | Perioperative
Overall patient satisfaction | After hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Tedore, M.D., Principal Investigator — New York Presbyterian Hospital Weill Cornell Medical Center
Locations (1):
- New York Presbyterian Hospital Weill Cornell Medical Center, New York, New York, United States

REFERENCES:
- [Background] Pusch F, Freitag H, Weinstabl C, Obwegeser R, Huber E, Wildling E. Single-injection paravertebral block compared to general anaesthesia in breast surgery. Acta Anaesthesiol Scand. 1999 Aug;43(7):770-4. doi: 10.1034/j.1399-6576.1999.430714.x. PMID 10456819
- [Background] McCartney CJ, Brull R, Chan VW, Katz J, Abbas S, Graham B, Nova H, Rawson R, Anastakis DJ, von Schroeder H. Early but no long-term benefit of regional compared with general anesthesia for ambulatory hand surgery. Anesthesiology. 2004 Aug;101(2):461-7. doi: 10.1097/00000542-200408000-00028. PMID 15277930
- [Background] Coveney E, Weltz CR, Greengrass R, Iglehart JD, Leight GS, Steele SM, Lyerly HK. Use of paravertebral block anesthesia in the surgical management of breast cancer: experience in 156 cases. Ann Surg. 1998 Apr;227(4):496-501. doi: 10.1097/00000658-199804000-00008. PMID 9563536
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Karmakar MK, Booker PD, Franks R. Bilateral continuous paravertebral block used for postoperative analgesia in an infant having bilateral thoracotomy. Paediatr Anaesth. 1997;7(6):469-71. doi: 10.1046/j.1460-9592.1997.d01-118.x. PMID 9365974
- [Background] Richardson J, Vowden P, Sabanathan S. Bilateral paravertebral analgesia for major abdominal vascular surgery: a preliminary report. Anaesthesia. 1995 Nov;50(11):995-8. doi: 10.1111/j.1365-2044.1995.tb05939.x. PMID 8678263
- [Background] Wassef MR, Randazzo T, Ward W. The paravertebral nerve root block for inguinal herniorrhaphy--a comparison with the field block approach. Reg Anesth Pain Med. 1998 Sep-Oct;23(5):451-6. doi: 10.1016/s1098-7339(98)90026-8. PMID 9773696
- [Background] Eason MJ, Wyatt R. Paravertebral thoracic block-a reappraisal. Anaesthesia. 1979 Jul-Aug;34(7):638-42. doi: 10.1111/j.1365-2044.1979.tb06363.x. PMID 517716
- [Background] Gilbert J, Hultman J. Thoracic paravertebral block: a method of pain control. Acta Anaesthesiol Scand. 1989 Feb;33(2):142-5. doi: 10.1111/j.1399-6576.1989.tb02877.x. PMID 2922982
- [Background] Cheema SP, Ilsley D, Richardson J, Sabanathan S. A thermographic study of paravertebral analgesia. Anaesthesia. 1995 Feb;50(2):118-21. doi: 10.1111/j.1365-2044.1995.tb15092.x. PMID 7710020
- [Background] Terheggen MA, Wille F, Borel Rinkes IH, Ionescu TI, Knape JT. Paravertebral blockade for minor breast surgery. Anesth Analg. 2002 Feb;94(2):355-9, table of contents. doi: 10.1097/00000539-200202000-00023. PMID 11812698
- [Background] Evans PJ, Lloyd JW, Wood GJ. Accidental intrathecal injection of bupivacaine and dextran. Anaesthesia. 1981 Jul;36(7):685-7. doi: 10.1111/j.1365-2044.1981.tb08781.x. PMID 6168207
- [Background] Lonnqvist PA, MacKenzie J, Soni AK, Conacher ID. Paravertebral blockade. Failure rate and complications. Anaesthesia. 1995 Sep;50(9):813-5. doi: 10.1111/j.1365-2044.1995.tb06148.x. PMID 7573876
- [Background] Chan VWS, Perlas A, Rawson R, Odukoya O. Ultrasound-guided supraclavicular brachial plexus block. Anesth Analg. 2003 Nov;97(5):1514-1517. doi: 10.1213/01.ANE.0000062519.61520.14. PMID 14570677
- [Background] Marhofer P, Sitzwohl C, Greher M, Kapral S. Ultrasound guidance for infraclavicular brachial plexus anaesthesia in children. Anaesthesia. 2004 Jul;59(7):642-6. doi: 10.1111/j.1365-2044.2004.03669.x. PMID 15200537
- [Background] Sandhu NS, Manne JS, Medabalmi PK, Capan LM. Sonographically guided infraclavicular brachial plexus block in adults: a retrospective analysis of 1146 cases. J Ultrasound Med. 2006 Dec;25(12):1555-61. doi: 10.7863/jum.2006.25.12.1555. PMID 17121950
- [Background] Pusch F, Wildling E, Klimscha W, Weinstabl C. Sonographic measurement of needle insertion depth in paravertebral blocks in women. Br J Anaesth. 2000 Dec;85(6):841-3. doi: 10.1093/bja/85.6.841. PMID 11732516
- [Background] Greengrass R, O'Brien F, Lyerly K, Hardman D, Gleason D, D'Ercole F, Steele S. Paravertebral block for breast cancer surgery. Can J Anaesth. 1996 Aug;43(8):858-61. doi: 10.1007/BF03013039. PMID 8840066
- [Background] Weltz CR, Greengrass RA, Lyerly HK. Ambulatory surgical management of breast carcinoma using paravertebral block. Ann Surg. 1995 Jul;222(1):19-26. doi: 10.1097/00000658-199507000-00004. PMID 7618963
- [Background] Najarian MM, Johnson JM, Landercasper J, Havlik P, Lambert PJ, McCarthy D. Paravertebral block: an alternative to general anesthesia in breast cancer surgery. Am Surg. 2003 Mar;69(3):213-8; discussion 218. PMID 12678477
- [Background] Karmakar MK. Thoracic paravertebral block. Anesthesiology. 2001 Sep;95(3):771-80. doi: 10.1097/00000542-200109000-00033. No abstract available. PMID 11575553
- [Derived] Chhabra A, Roy Chowdhury A, Prabhakar H, Subramaniam R, Arora MK, Srivastava A, Kalaivani M. Paravertebral anaesthesia with or without sedation versus general anaesthesia for women undergoing breast cancer surgery. Cochrane Database Syst Rev. 2021 Feb 25;2(2):CD012968. doi: 10.1002/14651858.CD012968.pub2. PMID 33629404